CLINICAL TRIAL: NCT03009266
Title: Ischemic Memory Imaging With MCE
Brief Title: Ischemic Memory Imaging With Myocardial Contrast Echocardiography
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jonathan R. Lindner, MD, Professor, Oregon Health and Science University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00016794
Record Dates: First submitted 2016-12-28; First posted 2017-01-04 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia | interventions — Sonazoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Normal controls (Experimental): Normal controls who will undergo dose-ranging studies to determine the optimal dose of phosphatidylserine-containing microbubbles that does not produce delayed myocardial opacification on myocardial contrast echocardiography (MCE).
  Interventions: Drug: Sonazoid
- Patients with ACS (Experimental): Subjects with ACS who have undergone primary percutaneous intervention in whom MCE with phosphatidylserine-containing microbubbles will be performed to determine whether the risk area can be detected and spatially defined.
  Interventions: Drug: Sonazoid

INTERVENTIONS:
Drug: Sonazoid — Myocardial contrast echocardiography ischemic memory imaging using intravenous administration of Sonazoid

SUMMARY:
The overall aim of this study is to determine whether non-invasive imaging with myocardial contrast echocardiography using can provide information on the presence and spatial extent of recent myocardial ischemia by non-invasive echocardiographic imaging.

ELIGIBILITY:
NORMAL CONTROL GROUP

Inclusion Criteria:

* Normal control individuals

Exclusion Criteria:

* History of cardiovascular disease (coronary artery disease, MI, peripheral artery disease)
* allergy to eggs or ultrasound contrast agents
* known or detected right to left shunt
* presence of a wall motion abnormality
* pregnancy

ACS GROUP

Inclusion Criteria:

* Patients with diagnosis of acute coronary syndrome with either unstable angina or non-ST-elevation MI
* Referred for primary percutaneous intervention
* At least 1 high risk features (ST changes, positive troponin, wall motion abnormality)

Exclusion Criteria:

* allergy to eggs or ultrasound contrast agents
* hemodynamic instability or shock
* known or detected right to left shunt
* pregnancy
* multivessel CAD requiring multivessel PCI

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-07-07 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Dose optimization | 3 months
  Dose ranging in normal controls to define highest dose of ultrasound contrast agent that does not produce delayed opacification from myocardial retention
Detection of Ischemia | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- OHSU, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Davidson BP, Hodovan J, Layoun ME, Golwala H, Zahr F, Lindner JR. Echocardiographic Ischemic Memory Molecular Imaging for Point-of-Care Detection of Myocardial Ischemia. J Am Coll Cardiol. 2021 Nov 16;78(20):1990-2000. doi: 10.1016/j.jacc.2021.08.068. PMID 34763776